CLINICAL TRIAL: NCT01236872
Title: The Acute Effect of Beetroot Juice on Circulating Nitrate and Nitrite Levels and Blood Pressure in Normotensives and Hypertensives
Brief Title: The Acute Effect of Beetroot Juice in Normal and Hypertensive Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University College, London (Other)
Responsible Party: Gerry Leonard, Joint Research and Development Office, BLT/QMUL
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 08/H0703/91 Acute
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-07

CONDITIONS: Hypertension
Keywords: Nitrate; Nitrite; Vegetable; Aortic stiffness
MeSH Terms: conditions — Hypertension | interventions — Water

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beetroot juice (Experimental): 250ml beetroot juice ingestion
  Interventions: Dietary Supplement: Beetroot juice
- Water (Placebo Comparator): 250ml low-nitrate water placebo
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Beetroot juice — 250ml once of beetroot juice
  Arms: Beetroot juice
Dietary Supplement: Water — 250ml once of low-nitrate mineral water
  Arms: Water

SUMMARY:
Inorganic nitrate can be converted to nitrite and thence nitric oxide in humans. Nitric oxide is normally produced by the inner lining of blood vessels and helps keep blood vessels open and therefore blood pressure lower. In subjects with high blood pressure, the inner lining of the blood vessels does not function adequately. The investigators wish to investigate whether elevating systemic levels of inorganic nitrate (through provision of dietary nitrate-rich vegetables) can elevate levels of nitrate/nitrite in hypertensive subjects, and whether this has a beneficial effect on blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and females between 18 and 85 years of age, inclusive.
2. To be eligible, female subjects will be required to state that they are not pregnant, and will not become pregnant during the course of the study.
3. Body mass index (BMI) between 18 and 40 kg/m2
4. A signed and dated written informed consent prior to admission to the study
5. The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
6. Grade 1 hypertensive SBP 140-159 or DBP 90-99 on no anti-hypertensives, no target organ damage (TOD), low cardiovascular disease (CVD) risk

Exclusion Criteria:

1. History of symptomatic coronary artery disease, stroke, or other known atherosclerotic disease.
2. History of chronic viral hepatitis (including presence of hepatitis B surface antigen or hepatitis C antibody), or other chronic hepatic disorders.
3. History of increased liver function tests (ALT, AST) due to acute or chronic liver conditions, 3x above the upper limit of normal or bilirubin 1.5x above the upper limit of normal at screening.
4. Renal impairment with creatinine clearance (eGFR) of <50 ml/min at screening.
5. Current poorly controlled diabetes mellitus, defined as HbA1c >10% at Screen.
6. Subjects with LDLc, >7.5 mmol/l. Fasting TG level >6mmol/l.
7. History of heart failure defined as NYHA class II - IV or those with known severe LV dysfunction (EF<30%) regardless of symptomatic status
8. History of malignancy within the past 5 years, other than non-melanoma skin cancer.
9. Current life-threatening condition other than vascular disease (e.g., very severe chronic airways disease, HIV positive, life-threatening arrhythmias) that may prevent a subject from completing the study.
10. Alcohol or drug abuse within the past 6 months.
11. Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is the longer) preceding the first dose of study medication.
12. Subjects who will commence or who are likely to commence treatment with non-steroidal anti-inflammatory drugs (NSAIDs) (other than aspirin), from screening until study completion.
13. Any non-stable dosing of ongoing medication regimens throughout the study trial.
14. The subject has a three month prior history of regular alcohol consumption exceeding an average weekly intake of > 28 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 21 units (or an average daily intake of greater than 2 units) for females. 1 unit is equivalent to a halfpint (284mL) of beer/lager; 25mL measure of spirits or 125mL of wine; or a positive alcohol breath test at the screening visit
15. A positive urine test for drugs of abuse (not related to known medications the subject is taking, ie, codeine for pain management) or alcohol at screening or prior to study medication administration.
16. Any other subject whom the Investigator deems unsuitable for the study (e.g., due to either medical reasons, laboratory abnormalities, expected study medication noncompliance, or subject's unwillingness to comply with all study-related study procedures).
17. Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with chronic inflammation (e.g. Inflammatory Bowel Disease).
18. Subjects with any acute infection, or significant trauma (burns, fractures).
19. Subjects who have donated more than 500 mL of blood within 56 days prior to the initiation of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in circulating nitrate/nitrite/cGMP levels | 24 hours

SECONDARY OUTCOMES:
Changes in blood pressure | 24 hours
arterial stiffness | 3hours
  pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahluwalia, Principal Investigator — QMUL
Locations (1):
- Queen Mary University London, London, United Kingdom

REFERENCES:
- [Background] Kapil V, Milsom AB, Okorie M, Maleki-Toyserkani S, Akram F, Rehman F, Arghandawi S, Pearl V, Benjamin N, Loukogeorgakis S, Macallister R, Hobbs AJ, Webb AJ, Ahluwalia A. Inorganic nitrate supplementation lowers blood pressure in humans: role for nitrite-derived NO. Hypertension. 2010 Aug;56(2):274-81. doi: 10.1161/HYPERTENSIONAHA.110.153536. Epub 2010 Jun 28. PMID 20585108
- [Background] Webb AJ, Patel N, Loukogeorgakis S, Okorie M, Aboud Z, Misra S, Rashid R, Miall P, Deanfield J, Benjamin N, MacAllister R, Hobbs AJ, Ahluwalia A. Acute blood pressure lowering, vasoprotective, and antiplatelet properties of dietary nitrate via bioconversion to nitrite. Hypertension. 2008 Mar;51(3):784-90. doi: 10.1161/HYPERTENSIONAHA.107.103523. Epub 2008 Feb 4. PMID 18250365